CLINICAL TRIAL: NCT04078685
Title: Contact-Force-Sensing-Based Radiofrequency Catheter Ablation in Paroxysmal Supraventricular Tachycardias: a Randomized Controlled Trial
Brief Title: Contact-Force-Sensing-Based Radiofrequency Catheter Ablation in Paroxysmal Supraventricular Tachycardias
Acronym: COBRA-PATH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Tamás Géczy, Cardiologist, Erasmus Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL62017.078.17
Record Dates: First submitted 2019-09-02; First posted 2019-09-06 (Actual); Last update posted 2020-09-03 (Actual); Status verified 2020-09

CONDITIONS: Tachycardia; Paroxysmal, Supraventricular; Tachycardia, Supraventricular
MeSH Terms: conditions — Tachycardia, Ventricular; Tachycardia, Supraventricular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CONVENTIONAL group (Active Comparator): Patients with supraventricular tachycardia treated with radiofrequency ablation using a standard (non-contact-force sensing) ablation catheter
  Interventions: Procedure: Standard catheter ablation
- CONTACT-FORCE group (Experimental): Patients with supraventricular tachycardia treated with radiofrequency ablation using a Contact-Force-sensing ablation catheter
  Interventions: Procedure: Contact Force-sensing-based catheter ablation

INTERVENTIONS:
Procedure: Standard catheter ablation — Radiofrequency catheter ablation using a standard ablation catheters: not equipped with contact-force sensing
  Arms: CONVENTIONAL group
Procedure: Contact Force-sensing-based catheter ablation — Radiofrequency catheter ablation using a Contact-Force-sensing ablation catheter
  Arms: CONTACT-FORCE group

SUMMARY:
The aim of this single-center prospective randomized controlled trial is to assess the superiority of contact-force-(CF)-sensing-based approach compared to conventional (non-CF-sensing) approach in the catheter ablation of PSVTs, and to investigate the safety of open-irrigated, contact-force-sensing ablation catheters (used in a "non-irrigated" mode) in these procedures.

DETAILED DESCRIPTION:
Rationale:

Multiple studies have demonstrated the importance of adequate catheter-tissue contact in the creation of effective lesions during radiofrequency catheter ablation. The development of contact-force(CF)-sensing catheters have contributed significantly to improve clinical outcomes in atrial fibrillation 3-18. However CF-sensing technology is not used in the ablation of paroxysmal supraventricular tachycardia. Although PSVT ablation with the conventional approach (non-irrigated, non-CF-sensing catheters) is considered a relatively low-risk procedure with fairly high success rate (short-and long-term) 1,2,19, we hypothesize that contact-force sensing can further improve the outcomes of these procedures. Based on the results of studies on atrial fibrillation ablation (mentioned above) we believe that CF-sensing could similarly improve such important parameters as radiofrequency (RF) application number/time, total procedure time, and fluoroscopy time in cases of PSVT ablations, as well. In addition CF-sensing could also further improve acute success/recurrence rates of PSVT ablation, and might also be capable to further diminish complication risk.

Primary Objective:

The primary objective of the present study is to demonstrate the superiority of contact-force-sensing in the ablation of AVNRT and WPW-AVRT as assessed by the improvement in the number and duration of radiofrequency applications compared with the conventional ablation approach.

Secondary Objective:

Secondary objectives of the study are the followings:

* to demonstrate that contact-force-sensing catheters are superior in terms of total procedure duration and fluoroscopy times in the case of AVNRT/WPW-AVRT ablation.
* to show that the use of contact-force sensing catheters is non-inferior to conventional catheters (without contact-force-sensing) in terms of acute/long-term procedural success and procedural safety (major/minor complication rate) of AVNRT/WPW-AVRT ablations.

Study population:

All patients above 18 years without structural heart disease being referred for electrophysiological study and potential treatment with radiofrequency catheter ablation of atrioventricular nodal reentrant tachycardia (AVNRT) and atrioventricular reentrant tachycardia (AVRT) with manifest (WPW syndrome) or concealed accessory pathways.

Intervention:

One group undergoes manual ablation using standard non-irrigated ablation catheters and the other group undergoes manual ablation with an open-irrigated ablation catheter equipped with CF- sensing (and utilized in a non-irrigated mode during ablation)

Main study parameters/endpoints:

The main study endpoint is the difference in RF application number during the procedures of AVNRT/WPW-AVRT ablation; secondary endpoints are differences in RF application rate, acute success rate, long-term recurrence rate (1 year) major/minor complication rate, and total procedure/fluoroscopy time.

ELIGIBILITY:
Inclusion Criteria:

* Referral for electrophysiology study because of pre-excitation on 12-lead surface ECG and/or documented (or suspected) symptomatic PSVT
* Identification of AVNRT or WPW-AVRT (with manifest or concealed accessory pathway) during standard EP study
* Verbal consent to continue with ablation therapy
* Informed written consent to be included in the study

Exclusion Criteria:

* evidence of structural heart disease and/or myocardial ischemia
* pregnancy (and lack of exclusion of potential pregnancy)
* age below 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2018-06-12 (Actual); Primary Completion 2020-03-09 (Actual); Study Completion 2021-03-20 (Estimated)

PRIMARY OUTCOMES:
Number of radiofrequency applications | From the beginning till the end of the ablation procedure
  The number of radiofrequency applications during the ablation procedures of AVNRT and WPW-AVRT

SECONDARY OUTCOMES:
Overall duration of radiofrequency applications | From the beginning till the end of the ablation procedure
  total of time spend from the beginning till the end of the ablation procedure
Long-term procedural success | At 12 months
  Free from recurrence of pre-excitation or the same clinical type of paroxysmal supraventricular tachycardia (AVNRT or AVRT)
Acute procedural success/failure | at the end of the ablation procedure
  non-inducibility of clinical arrhythmia verified at the end of the standard EP study
Fluoroscopy time | From the beginning till the end of the ablation procedure
  total time for fluoroscopy time
Total duration of procedure | From the beginning till the end of the ablation procedure
  total time for duration of the procedure
(Serious) Adverse Events | Till 12 months
  all reported SAEs
Time to recurrence of AVNRT/WPW-AVRT | up till 12 months
  if recurrence of AVNRT/WPW-AVRT, time to recurrence

CONTACTS AND LOCATIONS:
Overall Officials: Tamas Szili-Torok, MD, PhD, Principal Investigator — Erasmus Medical Center
Locations (1):
- Erasmus MC, Rotterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ullah W, Hunter RJ, Haldar S, McLean A, Dhinoja M, Sporton S, Earley MJ, Lorgat F, Wong T, Schilling RJ. Comparison of robotic and manual persistent AF ablation using catheter contact force sensing: an international multicenter registry study. Pacing Clin Electrophysiol. 2014 Nov;37(11):1427-35. doi: 10.1111/pace.12501. Epub 2014 Sep 15. PMID 25220575
- [Background] Gerstenfeld EP. Contact force-sensing catheters: evolution or revolution in catheter ablation technology? Circ Arrhythm Electrophysiol. 2014 Feb;7(1):5-6. doi: 10.1161/CIRCEP.114.001424. No abstract available. PMID 24550405
- [Background] Shurrab M, Di Biase L, Briceno DF, Kaoutskaia A, Haj-Yahia S, Newman D, Lashevsky I, Nakagawa H, Crystal E. Impact of Contact Force Technology on Atrial Fibrillation Ablation: A Meta-Analysis. J Am Heart Assoc. 2015 Sep 21;4(9):e002476. doi: 10.1161/JAHA.115.002476. PMID 26391136
- [Background] Kautzner J, Neuzil P, Lambert H, Peichl P, Petru J, Cihak R, Skoda J, Wichterle D, Wissner E, Yulzari A, Kuck KH. EFFICAS II: optimization of catheter contact force improves outcome of pulmonary vein isolation for paroxysmal atrial fibrillation. Europace. 2015 Aug;17(8):1229-35. doi: 10.1093/europace/euv057. Epub 2015 Jun 3. PMID 26041872
- [Background] Kimura M, Sasaki S, Owada S, Horiuchi D, Sasaki K, Itoh T, Ishida Y, Kinjo T, Tomita H, Okumura K. Comparison of lesion formation between contact force-guided and non-guided circumferential pulmonary vein isolation: a prospective, randomized study. Heart Rhythm. 2014 Jun;11(6):984-91. doi: 10.1016/j.hrthm.2014.03.019. Epub 2014 Mar 18. PMID 24657428
- [Background] Kuck KH, Reddy VY, Schmidt B, Natale A, Neuzil P, Saoudi N, Kautzner J, Herrera C, Hindricks G, Jais P, Nakagawa H, Lambert H, Shah DC. A novel radiofrequency ablation catheter using contact force sensing: Toccata study. Heart Rhythm. 2012 Jan;9(1):18-23. doi: 10.1016/j.hrthm.2011.08.021. Epub 2011 Aug 26. PMID 21872560
- [Background] Martinek M, Lemes C, Sigmund E, Derndorfer M, Aichinger J, Winter S, Nesser HJ, Purerfellner H. Clinical impact of an open-irrigated radiofrequency catheter with direct force measurement on atrial fibrillation ablation. Pacing Clin Electrophysiol. 2012 Nov;35(11):1312-8. doi: 10.1111/j.1540-8159.2012.03503.x. Epub 2012 Sep 4. PMID 22946636
- [Background] Natale A, Reddy VY, Monir G, Wilber DJ, Lindsay BD, McElderry HT, Kantipudi C, Mansour MC, Melby DP, Packer DL, Nakagawa H, Zhang B, Stagg RB, Boo LM, Marchlinski FE. Paroxysmal AF catheter ablation with a contact force sensing catheter: results of the prospective, multicenter SMART-AF trial. J Am Coll Cardiol. 2014 Aug 19;64(7):647-56. doi: 10.1016/j.jacc.2014.04.072. PMID 25125294
- [Derived] Geczy T, Ramdat Misier NL, Szili-Torok T. Contact-Force-Sensing-Based Radiofrequency Catheter Ablation in Paroxysmal Supraventricular Tachycardias (COBRA-PATH): a randomized controlled trial. Trials. 2020 Apr 9;21(1):321. doi: 10.1186/s13063-020-4219-1. PMID 32272969